CLINICAL TRIAL: NCT06335277
Title: Total Body Irradiation Treatments for Patients Treated at European Institute of Oncology
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 0727
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Leukemia; Leukemia, Chronic; Leukemia, Acute; Lymphoma; Aplastic Anemia
MeSH Terms: conditions — Leukemia; Bronchiolitis Obliterans Syndrome; Lymphoma; Anemia, Aplastic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total Body Irradiation (TBI): Patients treated at European Institute of Oncology with Total Body Irradiation (TBI)

SUMMARY:
Patients eligible undergoing total body irradiation as candidates for bone marrow or peripheral stem cell transplant.

DETAILED DESCRIPTION:
Total Body Irradiation (TBI) is an oncological radiotherapy technique that has been used for several decades in patients undergoing bone marrow or peripheral stem cell transplantation.

The role of TBI is:

To suppress the recipient's immune system to prevent rejection of the donor's bone marrow, whether familial or non-familial.

To eradicate residual neoplastic cells following chemotherapy treatments.

TBI is typically employed in both neoplastic and non-neoplastic disorders affecting blood cell elements (e.g., acute and chronic leukemias, aplastic anemia, lymphomas, etc.), as well as other conditions such as neuroblastoma, Ewing's tumor, and pediatric sarcomas with a poor prognosis.

Treatment choice is usually established following multidisciplinary discussions, based on disease characteristics and stage, concurrent pathologies and pharmacological treatments, patient preferences, and functional aspects. Data collection related to radiotherapy plays a crucial role in understanding various clinical aspects of the treatment itself. The availability of data from an increasing number of patients will allow the identification of clinical situations or technical parameters of radiotherapy correlated with treatment tolerance and effectiveness, aiming to identify the best treatment for these oncological pathologies.

This project aims to collect data related to total body irradiation treatments for scientific dissemination with the goal of establishing the basis for evaluating achieved results over time and deriving from these elements useful for guiding the most effective treatment strategies and appropriate operational protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing total body irradiation as candidates for bone marrow or peripheral stem cell transplantation.
2. Signed informed consent

Exclusion Criteria:

* Patients who do not undergo total body irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at European Institute of Oncology with Total Body Irradiation (TBI)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5 years
  Number of patients death
Disease free survival | 5 years
  Number of oncological event (local recurrence, distant metastasis, other primary tumor)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Alicja Jereczek, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy